CLINICAL TRIAL: NCT06108583
Title: Evaluation of the Effectiveness of a Mixed (Multifamily Group) Psychological Intervention Program for Children With Autism Spectrum Disorder and Feeding Difficulties (ASD+FD)
Brief Title: Evaluation of the Effect of a Psychological Program for Children With Autism Spectrum Disorder and Feeding Difficulties
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Fundació Sant Joan de Déu (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: PIC-151-17
Record Dates: First submitted 2023-10-25; First posted 2023-10-31 (Actual); Last update posted 2025-04-27 (Actual); Status verified 2025-04

CONDITIONS: Autism Spectrum Disorder
Keywords: Autism; Feeding difficulties; Clinical trial; Intervention
MeSH Terms: conditions — Autism Spectrum Disorder; Autistic Disorder

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Experimental group (Experimental): The experimental group received intervention with TEAlimento program. The intervention combines parent training in both group and individual sessions, as well as group sessions with children.
  The program is made up of 12 sessions, focuses on parent training and uses video-modeling. Additionally, a post-group individual session is conducted three months after the intervention. Sessions are held weekly, combining group (1.5 h) with individual (1 h) sessions. During group sessions, caregivers attend a parent training session, which is focused on teaching strategies based on the principles of behavior intervention and specific techniques related to eating. Simultaneously, children attend a group session in a separate room to target sensory issues and receive oral-facial stimulation. Individual sessions are held only with caregivers in order to individualize strategies to target the needs of each child. Each group includes from 3 to 5 participants.
  Interventions: Behavioral: TEAlimento : a multicomponent parent training behavioral program to treat feeding difficulties in children with Autism Spectrum Disorder
- Control group (No Intervention): The control group included participants in a waiting list. These families completed questionnaires at baseline and three months later (same time points as the experimental group), but they did not receive intervention during this period.
  Intervention was provided afterwards, but data after participating in the program was not included in this study.

INTERVENTIONS:
Behavioral: TEAlimento : a multicomponent parent training behavioral program to treat feeding difficulties in children with Autism Spectrum Disorder — The program focuses on parent training. Additionally, intervention on sensory integration is implemented directly with children. The program is made up of 12 sessions, which are held weekly, combining group (1.5 hour parent training and child sensory desensitization) with individual sessions. Parent training group sessions (1,3,4,5,7,8), are focused on teaching strategies based on the principles of behavior intervention and specific techniques related to eating. Strategies involve functional behavioral assessment, antecedent-based interventions, extinction of disruptive behaviors, positive reinforcement, modeling and visual supports. Additionally, parents were trained in methods of introducing new foods, such as modifying food presentation or textures. Simultaneously, children attend a group session in a separate room to target sensory issues and receive oral-facial stimulation. Individual sessions (2,6,9) are focused on specific characteristics of each child.
  Arms: Experimental group

SUMMARY:
Feeding difficulties are frequent in children with Autism Spectrum Disorder (ASD). The main goal of this project was to develop TEAlimento, a behavioral program for children ages 3-8 with ASD and feeding difficulties. The intervention combines parent training in group and individual sessions, as well as group sessions with children. The second goal was to conduct a pilot study to evaluate the effect of the program.

It was hypothesized that the intervention would decrease food rejection and disruptive behavior during meals, as well as increase the number of foods tried. A decrease in parent stress was also expected.

DETAILED DESCRIPTION:
Feeding difficulties are frequent in children with Autism Spectrum Disorder (ASD). The first goal was to develop TEAlimento, a behavioral program for children ages 3-8 with ASD and feeding difficulties. The second goal was to conduct a pilot study to evaluate the effect of the program.

Design A randomized waitlist -controlled clinical trial was designed to evaluate the effect of the program. The study ompared the intervention condition at two time points: baseline and 3 months later (our intervention program consisted of 12 sessions with a frequency of one session per week).

Initial effectivity data will be evaluated through the following specific indicators: limited variety of food, food rejection, disturbing behavior during meals and parent stress. Questionnaires to assess eating behaviors and parent stress will be administered before and after the intervention. Additionally, the number of new foods and food categories accepted after the intervention will be quantified. It was hypothesized that the intervention would decrease food rejection and disruptive behavior during meals, as well as increase the number of foods tried. A decrease in parent stress was also expected.

After approval by the review board of the Research and Ethics Committee of the Hospital, participants were recruited by psychologists and psychiatrists from a Multidisciplinary Unit for Autism Spectrum Disorder of a Child and Adolescent Mental Health Service, in accordance with the 2000 Helsinki Declaration.

Instruments

Characterization measures In order to confirm the diagnosis of autism spectrum disorder, clinical interviews were conducted with parents and the Autism Diagnostic Observational Schedule-2 was administered to all participants. To be included in the study, a score above the ADOS-2 cut-off point was requested. Intellectual ability was measured with the Weschler Preschool and Primary Scale of Intelligence IV or the Weschler Intelligence Scale for Children V, according to age. Adaptative functioning was measured with the Vineland Scale-2. In order to obtain specific information related to the child's food history, an ad hoc food history record was also filled with parents.

Outcome measures

In order to obtain preliminary data of the effect of the program, different instruments were administered before and after the intervention:

* Parenting Stress Index, short version (PSI).
* Brief Assessment of Mealtime Behavior In Children (BAMBIC).
* Qualitative questionnaire. To collect information about the amount of new accepted foods and new categories of food accepted before and after the intervention, the investigators conducted interviews with parents at the beginning of each session and filled a specific food questionnaire (ad hoc/qualitative data)., with different categories of food: dairy products (milk, cheese); eggs, meat and fish; vegetables (green beans, tomatoes, lettuce); fruit (apple, banana, almonds, peanuts); beans (lentils, beans) and cereals (rice, bread); pastry (croissants, cakes, chocolate); miscellany (mayonnaise, spicy, fritters, snacks); and drinks (juices, soft drinks, water). Additionally, the questionnaire registered the tastes that the child accepted (salty, sweet, acid or sour) and the accepted colors for meals (red, green, white).

Procedures

After receiving information about the study, parents provided signed consent. Included participants were invited to participate in the TEAlimento program, a behavioral program to treat feeding difficulties in children with ASD between 3 and 8 years of age. The intervention combines parent training in both group and individual sessions, as well as group sessions with children. The program includes behavioral techniques, such as functional behavioral assessment, antecedent-based interventions, extinction of disruptive behaviors during meals, positive reinforcement (praise, access to toys or engaging in preferred activities), modeling and visual supports. Additionally, parents were trained in methods of introducing new foods, such as modifying the bite size, food presentation or food texture. Parents also received information about recommended mealtime routines, such as structured time tables and calm environment during meals.

The program focuses on parent training and uses video-modeling. The program is made up of 12 intervention sessions, divided into three phases: functional assessment (3 sessions), direct intervention (8 sessions), and closing (1 session). In addition, this structure is complemented by an initial telephone evaluation and a pre-group group session with the caregiver. Additionally, a post-group individual session with the caregiver is conducted three months after the intervention.

Sessions are held weekly, combining group (1.5 h) with individual (1 h) sessions. During group sessions (sessions 1,3,4,5,7,8), caregivers attend a parent training session. Parent training is focused on teaching strategies based on the principles of behavior intervention, management of contingencies and specific techniques related to eating. Simultaneously, while parents receive this training, children attend a group session in a separate room to target sensory issues and receive oral-facial stimulation. Children work on sensory processing, playing with different types of sensory elements, trying to normalize their eating behavior and eating different kinds of food. Individual sessions (sessions 2,6,9) are held only with caregivers. These sessions are focused on specific characteristics and particular difficulties of each child, in order to individualize strategies to target the needs of each child.

For this study, each group included from 3 to 5 participants. Each group was conducted by either two psychologists or by one psychologist and a master degree student. The clinical team had large experience in interventions with ASD children. In order to ensure fidelity of implementation of the intervention, before each session, clinicians reviewed specific protocol instructions. By the end of each session, clinicians reviewed again the protocol, to ensure that the intervention was provided consistently as designed. Simultaneous group sessions with children were conducted by a mental health specialized nurse and the support of two master degree students.

Data Analysis The Statistical Package for the Social Sciences will be used for statistical analyses. Descriptive analyses will be conducted to characterize the sample. In order to evaluate whether there is a treatment effect on the feeding difficulties, a 2 X 2 (time x treatment group) ANOVA will be conducted for the following outcomes : limited variety of food, food rejection, disturbing behavior during meals, number of new foods and food category accepted and parent stress.

ELIGIBILITY:
Inclusion Criteria:

* age range between 3 and 8 years old
* confirmed diagnosis of cut-off at the Autism Diagnostic Observation Schedule-2 (ADOS-2, Lord et al., 2000)
* presence of significant feeding difficulties, defined as one or more of the following issues: significant food rejection, significant disruptive behavior at meals, significant selectivity based on type, texture, and presentation, and significant stress to family caused by these feeding difficulties.
* acquired oral-motor abilities to chew food
* accepts eating at least three foods (and a maximum of 20).

Exclusion Criteria:

* severe intellectual disability (intellectual or adaptive functioning below 35)
* severe behavioral problems
* medical risk situation that required more intensive intervention.

Ages: 3 Years to 8 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 30 (Estimated)
Dates: Start 2018-01-10 (Actual); Primary Completion 2026-12-31 (Estimated); Study Completion 2026-12-31 (Estimated)

PRIMARY OUTCOMES:
Change in Brief Assessment of Mealtime Behavior In Children (BAMBIC; Hendy et al. 2013). | Before and after intervention (12 weeks later)
  This questionnaire consists of 11 items that evaluate, on a 5-point Likert scale, three areas: limited variety, food refusal and disturbing behavior, in the last 6 months. Higher scores reflect more difficulties. The limited variety subscale assesses the child's willingness to try new foods or new types of preparation or textures. The food refusal subscale evaluates problem behaviors during meals, such as crying or closing his/her mouth tightly when food is presented. The disruptive behavior subscale includes items that assess aggressive behavior, self-injurious behaviors or disruptive conducts during meals, such as pushing or throwing utensils or food.

SECONDARY OUTCOMES:
Change in Parenting Stress Index, short version (PSI-SF; Abidin 1995). | Before and after intervention (12 weeks later)
  The PSI-SF includes three subscales, comprising 12 items each, rated from 1 to 5. The subscale Paternal Distress assesses the discomfort experienced by parents, such as poor sense of competence, lack of social support or depressive symptoms. The subscale Parent-Child Dysfunctional Interaction evaluates the degree in which the child meets the expectations that parents have and the reinforcement that the child offers to his/her parents. The subscale Difficult Child assesses the degree in which parents perceive how difficult it is to control their child, according to his/her behaviors. Finally, the instrument includes a total scale score, which is calculated by summing the three subscales' scores, ranging from 36 to 180. Scores of 90 or above may indicate a clinical level of stress.
Change in Qualitative questionnaire (ad hoc) | Before and after intervention (12 weeks later)
  To collect information about the amount of new accepted foods and new categories of food accepted before and after the intervention, we conducted interviews with parents at the beginning of each session and filled a specific food questionnaire (ad hoc/qualitative data)., with different categories of food: dairy products (milk, cheese); eggs, meat and fish; vegetables (green beans, tomatoes, lettuce); fruit (apple, banana, almonds, peanuts); beans (lentils, beans) and cereals (rice, bread); pastry (croissants, cakes, chocolate); miscellany (mayonnaise, spicy, fritters, snacks); and drinks (juices, soft drinks, water). Additionally, the questionnaire registered the tastes that the child accepted (salty, sweet, acid or sour) and the accepted colors for meals (red, green, white).

CONTACTS AND LOCATIONS:
Overall Officials: Maria A Mairena, PhD, Principal Investigator — Child and Adolescent Mental Health Research Group. Institut de Recerca Sant Joan de Déu. Spain
Locations (1):
- Department of Child and Adolescent Mental Health. Hospital Sant Joan de Déu, Esplugues de Llobregat, Barcelona, Spain

IPD SHARING:
Plan to Share IPD: No